CLINICAL TRIAL: NCT00872859
Title: The BREASTrial: Breast Reconstruction Evaluation Using Acellular Dermal Matrix as a Sling Trial
Brief Title: The BREASTrial:Breast Reconstruction Evaluation Using Acellular Dermal Matrix as a Sling Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jay Agarwal, Chief of the Division of Plastic Surgery, Associate Professor of Surgery, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26658
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer; Reconstructive Surgery
Keywords: Breast Cancer; Cancer of Breast; Reconstructive Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Alloderm

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Dermamatrix with radiation
  Interventions: Procedure: Implantation of Dermal Matrix substitute
- 2 (Experimental): Dermamatrix without radiation
  Interventions: Procedure: Implantation of Dermal Matrix substitute
- 3 (Experimental): Alloderm with radiation
  Interventions: Procedure: Implantation of Dermal Matrix substitute
- 4 (Experimental): Alloderm without radiation
  Interventions: Procedure: Implantation of Dermal Matrix substitute

INTERVENTIONS:
Procedure: Implantation of Dermal Matrix substitute — Dermal Matrix implanted in post mastectomy pts at time of mastectomy.
  Other Names: Dermamatrix; Alloderm; Dermal Matrix

SUMMARY:
Primary Hypothesis:

1. Alloderm and Dermamatrix have comparable complication rates when used for staged breast reconstruction

Secondary hypotheses:

1. The complication rates following staged breast reconstruction using Alloderm or Dermamatrix are higher if the patient requires radiation compared to those who do not require radiation.
2. Dermal matrix incorporation is not altered in patients requiring radiation compared to those who do not require radiation.
3. Dermal matrix incorporation is no different when comparing Alloderm and Dermamatrix

Specific aims:

1. Evaluate the complication rates in women undergoing staged breast reconstruction with acellular dermal matrix with or without radiation
2. Compare the complication rates between the two types of acellular dermal matrix
3. Evaluate the histologic characteristics of the dermal matrix exposed to radiation compared to that not exposed to radiation.
4. Compare the rates of incorporation of the dermal substance into surrounding tissues of those patients undergoing radiation to those not undergoing radiation

ELIGIBILITY:
Inclusion Criteria:

* Plan for immediate temporary breast reconstruction with tissue expander placement and acellular dermal matrix in patients undergoing mastectomy
* Female gender
* Age between 18 and 80
* Consent to participate in the study

Exclusion Criteria:

* Patients not undergoing breast reconstruction following mastectomy
* Patients undergoing delayed breast reconstruction following mastectomy
* Patients undergoing immediate definitive breast reconstruction after mastectomy
* Patients requiring definitive reconstruction within 3 months of immediate temporary breast reconstruction
* Medical debility precluding surgical treatment
* Prior breast or chest wall irradiation
* Pregnant patients
* Male gender

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Effects of radiation on acellular dermal matrix | four years

CONTACTS AND LOCATIONS:
Overall Officials: Jayant Agarwal, MD, Principal Investigator — University of Utah Hospital
Locations (1):
- University of Utah Hospital/ Huntsman Cancer Institute, Salt Lake City, Utah, United States